CLINICAL TRIAL: NCT02176317
Title: Autologous Umbilical Cord Blood Infusion for Children With Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: The Marcus Foundation (Other); PerkinElmer, Inc. (Industry)
Responsible Party: Principal Investigator, Joanne Kurtzberg, MD, Professor of Pediatrics, Duke University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00052449
Record Dates: First submitted 2014-06-16; First posted 2014-06-27 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; ASD; Umbilical cord blood; Autologous cord blood; cord blood
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous Umbilical Cord Blood (UCB) (Experimental): All participants will receive a single intravenous (into the vein) infusion of autologous umbilical cord blood cells.
  Interventions: Biological: Autologous Umbilical Cord Blood

INTERVENTIONS:
Biological: Autologous Umbilical Cord Blood — All participants will receive autologous umbilical cord blood cells with a pre-cryopreservation cell dose of 1-5 x 10^7 Total Nucleated Cells (TNC)/kilogram of subject body weight. The cells will be administered as a single intravenous (into the vein) infusion over 2 to 25 minutes

SUMMARY:
This study is a prospective phase 1 single-center trial designed to determine the safety of a single intravenous infusion of autologous umbilical cord blood in children with Autism Spectrum Disorder (ASD) and assess the feasibility of various outcome measures to determine which measure(s) can be used as primary and secondary endpoints for a future randomized phase 2 clinical trial. All subjects will receive infusion of cord blood cells at baseline with follow up assessments at 6 and 12 months.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopment disorder with early onset in life. Currently, available treatments for patients with ASD are supportive, but not curative. Umbilical cord blood (UCB) has been shown to lessen the clinical and radiographic impact of hypoxic brain injury and stroke in animal models and in infants with hypoxic ischemic encephalopathy. UCB also engrafts and differentiates in the brain, facilitating neural cell repair in animal models and human patients with inborn errors of metabolism undergoing allogeneic, unrelated donor UCB transplantation. Infusion of autologous UCB does not require immunosuppression and has been shown to be safe in young children with brain injuries such as cerebral palsy and stroke. In this study, the investigators hypothesize that infusion of a patient's own umbilical cord blood cells (UCB) can offer neural protection/repair in the brain and reduction of inflammation associated with this disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 24 months to ≤72months at the time of visit 1
2. Confirmed clinical DSM-5 diagnosis of Autism Spectrum Disorder using all three of the following measures:

   * Autism Diagnostic Observation Schedule - Toddler or Generic (ADOS)
   * Autism Diagnostic Interview-Revised (ADI-R)
   * DSM-5 checklist
3. IQ ≥ 35 on Stanford Binet Intelligence Scale or similar standardized test
4. Autologous umbilical cord blood available from a cord blood bank with a minimum total nucleated cell dose of ≥ 1 x 107 cells/kilogram of subject weight that meets acceptance criteria outlined in section 6.0 with confirmed HLA matching
5. Stable on current medications for at least 2 months prior to infusion of cord blood
6. Ability to travel to Duke University three times (0, 6, 12 mo.), parent/guardian able to participate in electronic communication tracking two times in the study and interim phone surveys every 3 months
7. Parental consent
8. Subject and parent/guardian must be English speaking

Exclusion Criteria:

1. Unwilling to commit to follow up for a year
2. History of prior cell therapy
3. Use of IVIG or other anti-inflammatory medications with the exception of NSAIDs
4. Medical records indicate that child has genetic or other syndromes such as fragile X, neurofibromatosis, Rett syndrome, tuberous sclerosis, PTEN mutation, cerebral palsy, cystic fibrosis, muscular dystrophy, Crohn's disease, or rheumatoid disease
5. Co-morbid condition that would influence child's performance on assessments.
6. Central Nervous System (CNS) infection
7. History of unstable epilepsy or uncontrolled seizure disorder, infantile spasms, Lennox Gastaut syndrome, Dravet syndrome
8. Known pathogenic copy number variation (CNV) (e.g. 16p11.2, 15q13.2, 2q13.3)
9. Significant sensory (i.e., deafness, blind) or motor impairment (CP) (if using Language Environment Analysis (LENA), no uncorrected hearing impairment)
10. Presence of obvious physical dysmorphology
11. Review of medical records indicates ASD diagnosis not likely or other serious complicating genetic or medical condition present
12. Impaired renal or liver function as determined by serum creatinine >1.5mg/dL and/or total bilirubin>1.3mg/dL
13. Clinically significant abnormalities in Complete Blood Count (CBC): Hemoglobin < 10.0 g/dL, White Blood Count (WBC) < 3.8 x 10e9, Platelets < 150x 10e9.
14. Known metabolic disorder, mitochondrial dysfunction
15. Uncontrolled infection, presence of or infection with HIV
16. Active malignancy
17. Macroencephaly or microencephaly ( >2 standard deviations in the relevant direction between head circumference and height)
18. Change in current stable use of psychoactive medications; as per parent report.

Ages: 24 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with non-serious and serious adverse events. | up to 12 months

SECONDARY OUTCOMES:
The primary efficacy measure will be change in the Vineland Adaptive Behavior Scale- II | up to 12 months

OTHER OUTCOMES:
Change in Pervasive Developmental Disorder- Behavior Inventory | up to 12 months
Change in Repetitive Behavior Scal | up to 12 months
Change in Sensory Experience Questionnaire | up to 12 months
Change in Behavior Assessment of Children | up to 12 months
Change in Autism Diagnostic Observation Scale | up to 12 months
Change in Clinical Global Impression- Severity and Improvement Scales | up to 12 months
Change in Stanford Binet Intelligence Scale or other standardized IQ test | up to 12 months
Change in frequency of child vocalization/ conversational turns | up to 12 months
Change in Expressive One-Word Picture Vocabulary Test | up to 12 months
Change in Preschool Age Psychiatric Assessment | up to 12 months
Change in Aberrant Behavior Checklist | up to 12 months
Prevalent and incident of GI symptoms | up to 12 months
Change in Parenting Stress Index | up to 12 months
Change in attention to social stimuli assessed via eye-tracking and electroencephalography (EEG) | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Simhal AK, Carpenter KLH, Nadeem S, Kurtzberg J, Song A, Tannenbaum A, Sapiro G, Dawson G. Measuring robustness of brain networks in autism spectrum disorder with Ricci curvature. Sci Rep. 2020 Jul 2;10(1):10819. doi: 10.1038/s41598-020-67474-9. PMID 32616759